CLINICAL TRIAL: NCT01550887
Title: Evaluation of Impulsivity on Cocaine and Crack Addicts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, JGalduroz, Dr., Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ANNA2011
Record Dates: First submitted 2011-12-12; First posted 2012-03-12 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Substance Dependence
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Impulsivity evaluation (No Intervention)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be performed on this study
  Other Names: No intervention will be performed on this study

SUMMARY:
This study main objective is investigating impulsivity on cocaine or crack addicts. The investigators main hypothesis is that different measures (such as scales or behavioral tasks, for example) of impulsivity may produce distinct outcomes, and they might also differ among cocaine (sniffed) and crack users. Thus, it would be of great value to compare such measures once these data are often interpreted as the same phenomenon.

DETAILED DESCRIPTION:
Drug dependence is characterized by a sum of cognitive, behavioral and physiological symptoms. Among these symptoms are the lack of control over ones own behavior and substance use even in face of significant issues related to it. Impulsivity (expressed as impulsive choice or fail on behavioral inhibition) is important in crucial phases of drug dependence development. Both behavioral and neurobiological studies have confirmed the association between impulsivity and addictive behaviors. Thus a high impulsivity level might have influence on patients' treatment. Even though, several questions on this matter remain unclear for humans, such as the differences on impulsivity between users of different forms of cocaine (either sniffed or smoked). This kind of difference could establish distinct ways of treatment and then enable developing better treatments for drug users. For this study it will be recruited 60 non-treated dependent patients, among them 30 cocaine users and 30 crack users. These individuals will be selected based on DSM-IV dependence criteria. The instruments used will be scales to measure compulsion and consumption of cocaine/crack, a pharmacological screening for psychotropic drugs and a cognitive evaluation. As impulsivity measures are Barratt Impulsivity Scale (BIS 11), a reward discounting questionnaire and a computer-based behavioral test on "ProgRef v3" software. For data analysis the impulsivity measures will be compared with the behavioral and cognitive instruments through the Pearson's correlation matrix. An ANOVA will be also performed to verify any differences between cocaine and crack dependents on the impulsivity and compulsion tests. When it is appropriate subsequent Newman-Keuls post-hoc test will be performed. Significance level adopted is 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-50 years old
* Cocaine/ Crack dependence criteria according to DSM-IV
* Have at least high school education level

Exclusion Criteria:

* Present dependence criteria for other drugs, except for Nicotine/tabacco
* Have any other psychiatric conditions

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2014-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Impulsive trait, as measured by different tests. | An expected average of 2 months
  To mesure "impulsive trait", will be used the Barratt Impulsivity Scale (BIS 11), the Reward Discounting Questionnaire and a computer-based Behavioral Test on "ProgRef v3" software.

CONTACTS AND LOCATIONS:
Overall Officials: José C Galduróz, PhD, Principal Investigator — Universidade Federal de São Paulo
Locations (1):
- UDED, São Paulo, São Paulo, Brazil